CLINICAL TRIAL: NCT04293107
Title: Using the Paediatric Gastroesophageal Reflux Disease Symptom and Quality of Life Questionnaire (PGSQ) in Children With Cerebral Palsy: a Preliminary Validation Study
Brief Title: Gastro-oesophageal Reflux and NeuroDisability (Cerebral Palsy) in CHILDren
Acronym: GRANDCHILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poole Hospital NHS Foundation Trust (Other)
Collaborators: British Society of Paediatric Gastroenterology, Hepatology and Nutrition (Unknown)
Responsible Party: Sponsor
Other Study IDs: GRANDCHILD v2.0
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; GORD; Pediatrics; GERD in Children; Quality of Life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Content Validity Testing: Cohort of 6 parents/carers of children with cerebral palsy and GORD, who will be interviewed regarding the content validity of the PGSQ when used to assess symptoms of GORD in children with cerebral palsy.
- Phase 2: Reliability (test-retest) Testing: Cohort of 20 parents/carers of children with cerebral palsy and GORD, who will review and complete the adapted version of the PGSQ (post Phase 1) at two time points, two weeks apart.

SUMMARY:
This study assesses the content validity of the PGSQ for parents/carer of children with cerebral palsy and GORD, including features such as readability, face validity and acceptability for completion. This will be done via 6 interviews, with the PGSQ being altered as identified as required. Reliability (test-retest) of the adapted version of the PGSQ being assessed with a sample of 20 parents/carers.

DETAILED DESCRIPTION:
Gastro-oesophageal reflux disease (GORD) is a common condition, where acid from the stomach leaks up into the oesophagus (food pipe) causing highly unpleasant symptoms and sometimes needing hospital admission. Children with cerebral palsy suffer from a poorly contracting food pipe (oesophageal dysmotility). As a result, GORD is more problematic in these children and more common; of the 8000 children with cerebral palsy aged 5-16 in the UK, around half suffer from reflux disease. This is treated with medicines or surgery. There is not an accurate measure of their symptoms, though there is a suitable questionnaire in well children (the PGSQ). National Institute for Health and Clinical Excellence (NICE) have recommended research to assess the effectiveness of medicines to treat GORD in these children (NG1 research recommendation). In the first phase, the investigators will ask 6 parents/carers their opinions about the PGSQ using qualitative interviews, and alter the PGSQ if needed; then in the second phase, ask 20 parents/carers about their child's symptoms to understand the reliability of the PGSQ at two time points 2 weeks apart (test-retest). The investigators won't do any invasive tests on the children but will ask parents about their opinions of their children taking part in pH-impedance monitoring, which is used to assess severity of GORD and may be useful in designing future studies.

ELIGIBILITY:
Inclusion Criteria:

* Parents or carers of children with cerebral palsy (GMFCS level III-V) with symptoms of GORD or on treatment for presumed GORD, aged between 2-16 years.

Exclusion Criteria:

* Children whose parent/carer are not able to support their participation in the study in the opinion of the investigator (e.g. language/communication issue, health, burden).

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents/carers of children (2-16 years) with cerebral palsy and GORD.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Valid modified Paediatric Gastroesophageal Reflux Disease Symptom and Quality of Life Questionnaire (PGSQ) | 1 day
  Qualitative feedback on whether the Paediatric Gastroesophageal Reflux Disease Symptom and Quality of Life Questionnaire (PGSQ) needs modification or is useful and appropriate for patents/carers of children with cerebral palsy and GORD.

SECONDARY OUTCOMES:
Phase 2: Reliability of modified Paediatric Gastroesophageal Reflux Disease Symptom and Quality of Life Questionnaire (PGSQ) | 2 weeks
  The difference in scores in the modified PGSQ performed twice, 2 weeks apart, compared with visual analogue symptom (VAS) scores to demonstrate test-retest reliability. VAS scores run from a scale of 0 (no symptoms) to 10 (severe symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Tighe, MRCPCH, Principal Investigator — University Hospitals Dorset NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Poole Hospital NHSFT, Poole, Dorset
  - Poole Hospital, Poole, Dorset

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleinman L, Nelson S, Kothari-Talwar S, Roberts L, Orenstein SR, Mody RR, Hassall E, Gold B, Revicki DA, Dabbous O. Development and psychometric evaluation of 2 age-stratified versions of the Pediatric GERD Symptom and Quality of Life Questionnaire. J Pediatr Gastroenterol Nutr. 2011 May;52(5):514-22. doi: 10.1097/MPG.0b013e318205970e. PMID 21464757